CLINICAL TRIAL: NCT04109339
Title: Effects of Oxytocin on Hemodynamics in Patients Undergoing Laparoscopic Myomectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20190501
Record Dates: First submitted 2019-08-15; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Oxytocin; Hemodynamic Monitoring; Laparoscopic Surgery
Keywords: Oxytocin; Hemodynamic; Myomectomy
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 with no oxytocin (No Intervention)
- group 2 with oxytocin 10 U IM + oxytocin 10 U IV (Experimental)
  Interventions: Drug: Oxytocin
- group 3 with oxytocin 20 U IM + oxytocin 0 U IV (Experimental)
  Interventions: Drug: Oxytocin
- group 4 with oxytocin 0 U IM + oxytocin 20 U IV (Experimental)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — During the laparoscopic hysteromyomectomia operation, different doses of oxytocin was used with different routs.
  Arms: group 2 with oxytocin 10 U IM + oxytocin 10 U IV; group 3 with oxytocin 20 U IM + oxytocin 0 U IV; group 4 with oxytocin 0 U IM + oxytocin 20 U IV

SUMMARY:
This project will study the effect of oxytocin on hemodynamics in patients undergoing laparoscopic myomectomy, and how to prevent and manage such hemodynamic changes effectively.It provides a reference for the rational use of oxytocin in clinical practice, which can not only effectively contract the uterus and reduce bleeding, but also reduce the influence on hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia for gynecological laparoscopic surgery,ASA I~III

Exclusion Criteria:

* Oxytocin use contraindications

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes of traditional hemodynamic parameters after oxytocin use during laparoscopic hysteromyomectomia. | "before induction", "before incision", "before oxytocin intramuscular injection", and "20 sec, 40 sec, 60 sec, 80 sec, 100 sec, 120 sec, 140 sec, 160 sec,180 sec after oxytocin intramuscular injection".
  Parameters including SBP, DBP, MAP (mmHg) were measured by a Mostcare hemodynamic monitor.
Changes of traditional hemodynamic parameters after oxytocin use during laparoscopic hysteromyomectomia. | "before induction", "before incision", "before oxytocin intramuscular injection", and "20 sec, 40 sec, 60 sec, 80 sec, 100 sec, 120 sec, 140 sec, 160 sec,180 sec after oxytocin intramuscular injection".
  HR (beats/min) was measured by a Mostcare hemodynamic monitor.
Changes of volume management parameters after oxytocin use during laparoscopic hysteromyomectomia. | "before induction", "before incision", "before oxytocin intramuscular injection", and "20 sec, 40 sec, 60 sec, 80 sec, 100 sec, 120 sec, 140 sec, 160 sec,180 sec after oxytocin intramuscular injection".
  SVV (%) was measured by a Mostcare hemodynamic monitor.
Changes of volume management parameters after oxytocin use during laparoscopic hysteromyomectomia. | "before induction", "before incision", "before oxytocin intramuscular injection", and "20 sec, 40 sec, 60 sec, 80 sec, 100 sec, 120 sec, 140 sec, 160 sec,180 sec after oxytocin intramuscular injection".
  SVRI (dynes-sec/cm-5) was measured by a Mostcare hemodynamic monitor.
Changes of volume management parameters after oxytocin use during laparoscopic hysteromyomectomia. | "before induction", "before incision", "before oxytocin intramuscular injection", and "20 sec, 40 sec, 60 sec, 80 sec, 100 sec, 120 sec, 140 sec, 160 sec,180 sec after oxytocin intramuscular injection".
  CI (l/min/m2) was measured by a Mostcare hemodynamic monitor.
Changes of volume management parameters after oxytocin use during laparoscopic hysteromyomectomia. | "before induction", "before incision", "before oxytocin intramuscular injection", and "20 sec, 40 sec, 60 sec, 80 sec, 100 sec, 120 sec, 140 sec, 160 sec,180 sec after oxytocin intramuscular injection".
  CO (l/min) was measured by a Mostcare hemodynamic monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China